CLINICAL TRIAL: NCT05957757
Title: RC48 Combined With Tislelizumab for Bladder Sparing Treatment in High-risk Non-muscular Invasive Bladder Cancer (NMIBC) With BCG Treatment Failure and HER2 Expression
Brief Title: RC48 Combined With Tislelizumab for Bladder Sparing Treatment in NMIBC With BCG Treatment Failure and HER2 Expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: RemeGen Co., Ltd. (Industry); BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-2022-021-B
Record Dates: First submitted 2023-05-12; First posted 2023-07-24 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Non-Muscle Invasive Bladder Cancer; HER2
Keywords: Non-Muscle Invasive Bladder Cancer; HER2 expression; BCG Failure; Unsuitable or refused to radical cystectomy
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — disitamab vedotin; tislelizumab

STUDY DESIGN:
Intervention Model Description: To study the safety and efficacy of RC48 combined with Tislelizumab in HER2 expression high grade non muscle invasive bladder cancer patients who failed BCG therapy and refused cystectomy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC48+Tislelizumab (Experimental): Approximately 20 subjects will be enrolled to evaluate the efficacy and safety of RC48 (RC48 2.0 mg/kg intravenously administered every two weeks) combined with Tislelizumab (Tislelizumab 200 mg intravenously administered every three weeks).
  Interventions: Drug: RC48; Drug: Tislelizumab

INTERVENTIONS:
Drug: RC48 — RC48 was scheduled to be administered at a dose of 2.0mg/kg every 2 weeks, with the first dose on day 1 of the first cycle.
  The drug is diluted with normal saline and administered by intravenous drip for one hour.
  Other Names: Disitamab Vedotin
Drug: Tislelizumab — Tislelizumab was administered at a dose of 200 mg every 3 weeks, with the first dose on day 1 of the first 21-day cycle.
  The drug is diluted with normal saline and administered by intravenous drip for one hour.

SUMMARY:
This is a prospective, open, single-center clinical study of anti-HER2-ADC combined with PD-1 monoclonal antibody for bladder sparing treatment in non-muscular invasive bladder cancer (NMIBC) patients with HER2-expressing. The study was conducted in accordance with the Good Clinical Practice (GCP). Approximately 20 subjects will be enrolled to evaluate the efficacy and safety of RC48 (RC48 2.0 mg/kg intravenously administered every two weeks) combined with Tislelizumab (Tislelizumab 200 mg intravenously administered every three weeks).

Subjects undergo Transurethral resection of bladder tumor (TURBT), imaging diagnosis and pre-treatment biological samples of blood, urine and biopsy tissue.

The study will include high-risk NMIBC patients who express HER2, fail after BCG treatment, but refuse to undergo cystectomy or do not meet the requirements for cystectomy.

Subjects will receive RC48 and Tislelizumab for two years. BI-DFS were evaluated by cystoscopy, histopathologic examination, laboratory examination, and imaging examination after treatment, and tumor efficacy was evaluated when clinical studies reached the number of subjects specified in the protocol for efficacy evaluation.

DETAILED DESCRIPTION:
For Non-muscle invasive bladder cancer (NMIBC), Transurethral resection of bladder tumor (TURBT) is the primary treatment. TURBT relapses within 12 months after surgery in 10% to 67% of patients, and postoperative bladder perfusion therapy (including chemotherapy and Immunotherapy) significantly reduces the recurrence rate. However, about 30%-40% of patients will relapse after BCG treatment. Radical cystectomy is the standard of care for patients who do not respond to BCG treatment and have high grade NMIBC. However, radical cystectomy has a high incidence of postoperative complications (up to 60%) and a negative impact on HRQoL. These complications occur even in high-volume centers of excellence, whether open or minimally invasive, and the mortality rate from the surgery itself is about 3%. Therefore, some patients refuse to undergo radical cystectomy. In addition, some patients are medically unfit for surgery due to age, functional status, American Society of Anesthesiologists classification, comorbiditions, body mass index, and other factors. Although penerubicin is the only bladder sparing drug approved by the U.S. Food and Drug Administration (FDA) for patients who are not suitable for or unwilling to undergo cystectomy, BCG refractory, and with CIS NMIBC, no legally marketed penerubicin drug is available in China. Therefore, new treatments are needed to prevent invasive bladder cancer from affecting the entire bladder.

In recent years, immunocheckpoint inhibitors represented by PD-1/PD-L1 have been proved to be a promising means of tumor immunotherapy, which has made a breakthrough in the treatment of advanced urothelial carcinoma, and become the main choice for the treatment of advanced urothelial carcinoma. Immunocheckpoint inhibitors also showed positive results in patients who did not respond to BCG treatment during perioperative and perioperative periods.Therefore, immunotherapy is expected to be an alternative bladder sparing therapy for high-risk NMIBC patients.The anti-HER2-ADC drug RC48 also achieved significant efficacy in HER2-overexpressed advanced urothelial carcinoma, and its combination with PD-1 monoclonal antibody Toripalimab was more effective in the first-line treatment of advanced metastatic urothelial carcinoma. Therefore, RC48 combined with PD-1 can be used as a potential treatment for bladder sparing in patients with NMIBC.

In NMIBC patients with HER2 expression, ADC drugs can target tumor cells and deliver cytotoxic drugs with greater safety than chemotherapy. In addition, the application of anti-HER2-ADC drugs combined with PD-1 in bladder sparing therapy is still lacking in experience and related studies. Therefore, we plan to conduct a study on bladder preservation therapy for patients with HER2-expressing NMIBC treated with ADC drugs combined with PD-1 monoclonal antibody, so as to preserve the bladder function of patients while controlling tumor recurrence and ensuring their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Histologically confirmed recurrent, non-muscle invasive bladder cancer;

   1. Histopathology: Patients with any variant urothelial cell carcinoma (UCC) (i.e., squamous and/or glandular epithelial differentiation UCC, UCC with micropapillary changes, nest variant UCC, plasmacytoid UCC, neuroendocrine UCC, and sarcomatoid UCC) were enrolled. The presence of any lymphatic infiltration (LVI) is considered evidence of high risk.
   2. Papillary carcinoma must be a high-risk disease defined as a high grade Ta/T1 lesion. In addition, subjects must have all visible tumors completely removed prior to initial administration of the study drug, as documented at baseline cystoscopy. Cytological results for high-grade urothelial carcinoma must be negative prior to initial administration of the investigational drug.
   3. CIS does not require complete excision, but must be completely excised with coexisting papillary carcinoma prior to enrollment and documented at baseline cystoscopy. Negative urine cytology for malignant cells is not required.
3. When BCG recurred after treatment, the presence of HER2 expression was detected by IHC in the pathology department of our hospital
4. BCG treatment failure included no response to BCG treatment and relapse after inadequate BCG treatment

   1. Subjects without response after adequate BCG treatment must meet at least one of the following criteria: 1) Persistent or recurrent simple CIS with or without recurrent Ta/T1 (non-invasive papillary carcinoma/tumor invasion of subepithelial connective tissue) disease within 12 months after completion of adequate BCG treatment; 2) Recurrent high-grade Ta/T1 disease occurred within 6 months after completion of adequate BCG treatment; 3) T1 high-grade disease was present at the first disease assessment after completion of a BCG induction course. Adequate BCG treatment (minimum treatment requirement) : at least 5 out of 6 full dose treatments were received during the initial induction course and at least 1 maintenance treatment within 6 months (one full dose per week and 2 out of 3 completed treatments); Or received at least 5 out of 6 full doses in the initial induction course and at least 2 out of 6 full doses in the second induction course.
   2. Relapse after inadequate BCG treatment: Subjects must meet the following criteria: Recurrence of high-grade Ta/T1 disease within 12 months of completion of BCG treatment (as defined below): Previous inadequate BCG treatment (minimum treatment requirement) included receiving at least 5 out of 6 full dose treatments during the initial induction course. Or received at least 5 out of 6 full dose treatments during the initial induction course and at least 1 maintenance treatment (once a week and 2 out of 3 completed treatments) within 6 months. One half or one third of the dose is allowed during maintenance treatment.
5. To refuse or be unsuitable for radical cystectomy
6. ECOG 0~1
7. The major organs are functioning normally, the following criteria are met:

(1) The blood routine examination criteria should meet (no blood transfusion and no treatment with granulocyte colony stimulating factor within 14 days before enrollment) : i. Absolute count of neutrophils (ANC) ≥1,000/mm3 ii. Platelet count ≥75,000/mm3 iii. Hemoglobin ≥ 8.0g /dL (2) Liver function: i. Total bilirubin ≤1.5× prescribed ULN or direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5×ULN ii. Upper limit of normal values (ULN) ≤2.5 times of alanine Aminotransferase (ALT) and aspartate Aminotransferase (AST) Note: ≤1.5× ULN (This criterion only applies to patients who have not received anticoagulant therapy; Patients receiving anticoagulant therapy should keep anticoagulants within therapeutic limits); (3) Kidney function: The Cockcroft-Gault formula was used to determine the creatinine clearance (CrCl) > 30 mL/min.

8. Subjects (or their legal representatives) must sign an informed consent form (ICF) indicating that they understand the purpose and procedures of the study and are willing to participate in the study; 9. Fertile women must have a negative pregnancy test result (beta-hCG) (urine or serum) within 7 days before the study drug is first administered.

Exclusion Criteria:

1. Confirmed by histology of muscular layer infiltration (T2 or higher level) bladder urothelial carcinoma.
2. Histopathological examination revealed any bladder small cell composition, pure, pure squamous cell carcinoma or simple squamous adenocarcinoma CIS;
3. Received other PD - 1 / PD - L1 inhibitor and/or HER2 inhibitor;
4. Active malignancies other than the disease being treated (i.e., disease progression within the last 24 months or requiring a change in treatment). Only the following special circumstances are allowed: i. Skin cancer that has been treated and completely cured within the last 24 months; ii. Adequately treated lobular carcinoma in situ (LCIS) and ductal CIS; iii. A history of local breast cancer and receiving antihormonal drugs or a history of local prostate cancer (N0M0) and receiving androgen blocking therapy.
5. History of uncontrolled cardiovascular disease, including: 1) any of the following in the past 3 months: unstable angina, myocardial infarction, ventricular fibrillation, toroidal ventricular tachycardia, cardiac arrest, or known congestive New York Heart Association Class III-IV heart failure, cerebrovascular accident, or transient ischemic attack; 2) Prolonged QTc interval confirmed by ECG evaluation during screening (Fridericia; QTc > 480 ms); 3) Pulmonary embolism or other venous thromboembolism within the past 2 months.
6. Pregnancy or lactation women;
7. Known human immunodeficiency virus (HIV) infection, unless the subjects in the past six months or longer had accepted the stability of antiretroviral therapy (art), and no opportunistic infections occurred in the past 6 months, and over the past six months the CD4 count of > 350;
8. Have evidence of active hepatitis B or hepatitis C infection (for example, a history of hepatitis C but hepatitis C virus polymerase chain reaction detection results and normal subjects of hepatitis B surface antigen antibody positive hepatitis B can groups);
9. Has yet to recover from past the toxic effects of anticancer therapy (except no clinical significance of toxic effects, such as hair loss, skin discoloration, neuropathy, and hearing impairment).
10. Wound healing delay, defined as the skin/decubitus ulcer, chronic leg ulcer, had known gastric ulcer or incision to heal.
11. 1 cycle day 1 major surgery within 4 weeks before (don't think TURBT belong to major surgery).
12. Other patients assessed by the investigator as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
2-yr Bladder-intact Disease-free Survival (BI-DFS) | Up to 24 months
  Defined by time from enrollment to the occurrence of one of the following events: first MIBC or regional lymph node recurrence, distant metastasis, or death

SECONDARY OUTCOMES:
Time to Progression (TTP) | Up to 24 months
  Defined by time from day of first treatment to first progression to higher grade or stage, including muscle-invasive disease or death from any cause.
Time to Deterioration (TTD) | Up to 24 months
  Defined by time from day of first treatment to first deterioration
Cystectomy Free Survival | Up to 24 months
  Defined by time from day of first treatment to radical cystectomy
Disease-Specific Survival (DSS) | Up to 24 months
  Defined by time from day of first treatment to invasive bladder cancer
Overall Survival (OS) | Up to 24 months
  Defined by time from day of first treatment to death
Percent of Patients With Complete Response (CR) | Up to 6 months
  CR is defined by negative cystoscopy, urine cytology, and bladder biopsies.
Recurrence Free Survival (RFS) | Up to 24 months
  Defined by time from day of first treatment to recurrent NMIBC based on cystoscopy, cytology and/or biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR